CLINICAL TRIAL: NCT06091215
Title: Combining Broad Based Light, Fractionated 1927 and Dual Wavelength 2940/1470 for Diffuse Pigmentation, Texture and Actinic Changes
Brief Title: Combining Broad Based Light (BBL), Fractionated 1927 (MOXI) and Dual Wavelength 2940/1470 (HALO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Sciton (Industry)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Principle Investigator, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1040
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Pigment Skin
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will receive 1-2 combination treatments.
Masking Description: PI will assess subject after a single treatment and decide if a second treatment is necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Single Treatment Arm (Active Comparator): Subjects will receive a single treatment of BBL/MOXI/HALO
  Interventions: Device: Sciton Joule System
- Double Treatment Arm (Active Comparator): Subjects will receive double treatment of BBL/MOXI/HALO 4-6 weeks apart.
  Interventions: Device: Sciton Joule System

INTERVENTIONS:
Device: Sciton Joule System — Sciton Joule System

SUMMARY:
This is a single-site, non-randomized, non-controlled study at UT Southwestern Medical Center at Dallas in the Department of Plastic Surgery. The study is designed to follow up to 15 consenting subjects who may receive up to 2 BBL/MOXI/HALO treatments under an IRB approved protocol.

DETAILED DESCRIPTION:
Subjects will receive 1-2 BBL/MOXI/HALO treatments. All 2nd treatments will be scheduled 4-8 weeks after the initial treatment to ensure the skin has enough time to recover. Overall assessments will be collected before the first treatment and at subsequent follow-up visits at 1 Month and 3 Months post final treatment. Identifiable full-face standard and close-up photography will be obtained and used to evaluate any changes. Subjects will also have photos obtained with the VISIA-CR Imaging System (Canfield Scientific, Parsippany, NJ). Quantitative analysis will be completed on the VISIA imaging system and be used to compare the effects of the treatments. Any improvements will be evaluated to pre-treatment assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults between 20-75 years of age
2. Fitzpatrick skin type 1-4
3. Individual deemed by the Investigator to benefit from skin resurfacing treatment(s)
4. Individuals willing to withhold aesthetic therapies that may potentially impact results to the treatment areas for the duration of the study
5. Women of childbearing potential:

   5.1. will be asked to agree to a pregnancy test before their screening visit in clinic 5.2. must use an acceptable method of birth control
   * Hormonal contraception (oral, injected, implanted, patch or vaginal ring)
   * Barrier method with spermicide: condom or occlusive cap with spermicidal foam/gel/cream/suppository
   * Intrauterine device (IUD)
   * Surgical Sterilization (e.gh., vasectomy, tubal occlusion, hysterectomy, bilateral salpingectomy/oophorectomy)
   * Abstinence from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject. Periodical abstinence and withdrawal methods are not acceptable forms of contraception.
6. Individuals who can read, speak, write and understand English and who are willing to provide written informed consent.
7. Individuals willing to sign a photography release with the understanding that their photos may be used during presentations at national conferences and/or published in journals
8. Individuals willing and able to cooperate with all study requirements for the duration of the study.

Exclusion Criteria:

1. Fitzpatrick skin type V-VI
2. Known allergies to general skin care products
3. Sensitivity to topical local anesthetic
4. Current or recent history of skin diseases:

   • Systemic granulomatous disease, either active or inactive, (e.g., Sarcoid, Wegener's, TB, etc) or connective tissue diseases (e.g., lupus, dermatomyositis, etc.)
5. Significant scars in the treatment area:

   * Severe or cystic and clinically significant acne or acne scars on the areas to be treated
   * Current or history of hypertrophic scarring or keloid scars
6. Tattoos in the area to be treated
7. Observable suntan, nevi, excessive hair, etc., or other dermal conditions that might influence study results on the face in the opinion of the Investigator
8. Individuals who currently have cancerous or pre-cancerous lesions in the area to be treated
9. Individuals with skin pathology and/or pre-existing dermatologic condition that the Investigator deems inappropriate for participation or could interfere with outcomes of the study, such as: psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, etc.
10. History of chronic drug or alcohol use
11. Recent aesthetic treatments:

    * <4 weeks of microdermabrasion or glycolic acid treatment to the treatment area or who plan to have this treatment during the study
    * <2 weeks of any type of injectable filler
    * <1 week of neurotoxin's
    * <6 months of ablative resurfacing laser treatments
    * <6 months of non-ablative, rejuvenative laser or light treatment
    * <3 months of chemical peels or dermabrasion
12. Use of the following prescription medications:

    * <6 weeks of Accutane or other systemic retinoids on the treatment area
    * <4 weeks of topical retinoids
    * <4 months of prescription strength lightening medications (e.g., hydroquinone, tretinoin, AHA, BHA, poly-hydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin)
    * <2 weeks of anti-wrinkle or skin lightening or topical systemic medication known to affect skin aging or dyschromia (e.g., alpha/beta/polyhydroxy acids, Vitamin C, soy, Q-10; hydroquinone, etc.,), TEGO, Cosmo C250, gigawhite, lemon juice extract (topically), or embilica extract
    * Antiplatelet agents/anticoagulant (Coumadin, Heparin, Plavix, chronic NSAID use)
    * Psychiatric drugs that would impair the subject from understanding protocol requirements or understanding and signing the ICF.
13. Individuals who are pregnant or planning to become pregnant during the course of the study
14. Immunocompromised individuals or those currently using immunosuppressive medications and/or radiation
15. Individuals with uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension, or hypothyroidism.
16. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures planned during the course of the study.
17. Individuals who, in the Investigator's opinion, have a history of poor cooperation, unreliability or noncompliance with medical treatment.
18. Individuals who are unable to understand instructions or give informed consent
19. Individuals who have physical or psychological conditions which, in the opinion of the Investigator, makes them unable to complete the study per protocol.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants- Single Treatment Group: Subjects will receive 1 BBL/MOXI/HALO treatments. Overall assessments will be collected before the first treatment and at subsequent follow-up visits at 1 Month and 3 Months post final treatment.
  Sciton Joule System: Sciton Joule System
- Healthy Participants- Double Treatment Group: Subjects will receive 2 BBL/MOXI/HALO treatments. All 2nd treatments will be scheduled 4-8 weeks after the initial treatment to ensure the skin has enough time to recover. Overall assessments will be collected before the first treatment and at subsequent follow-up visits at 1 Month and 3 Months post final treatment.
Period: Single treatment (4 weeks)
Arm/Group | Healthy Participants- Single Treatment Group | Healthy Participants- Double Treatment Group
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Double treatment (8 weeks)
Arm/Group | Healthy Participants- Single Treatment Group | Healthy Participants- Double Treatment Group
Started | 0 | 8
Completed | 0 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Treatment Arm | Double Treatment Arm | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Brown Spots at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall UV spots using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement
Time Frame: Baseline, 1 Month
Population: Analysis was focused on testing whether the effect of the treatment on each parameter differed
  The per-protocol (PP) population will be the primary population for all statistical analyses. The PP population will include all subjects who received treatment and completed the study in general accordance with the protocol. Only the data of completing subjects will be analyzed.
Measure: Median (Inter-Quartile Range); unit: count of spots
Groups:
- Single Treatment Arm: Quantitively assessment of intensity in overall brown spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of spots
  Front | 12.00 [-2.00 to 17.00]
  Left Oblique | 5.00 [-11.00 to 7.00]
  Nose | 0.00 [-3.00 to 1.00]
  Right Oblique | 5.00 [-11.00 to 5.00]

2. Primary Outcome: Change in Brown Spots at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of spots
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of spots
  Front | 8.00 [6.00 to 12.00]
  Left Oblique | .00 [-2.00 to 25.00]
  Nose | 3.00 [-1.00 to 5.00]
  Right Oblique | 9.00 [-2.00 to 25.00]

3. Primary Outcome: Change in Brown Spots at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of spots
Groups:
- Double Treatment Arm: Quantitively assessment of intensity in overall brown spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of spots
  Front | -2.00 [-14.00 to 0.50]
  Left Oblique | -3.50 [-9.00 to -0.50]
  Nose | -2.00 [-4.50 to -0.50]
  Right Oblique | -2.50 [-16.50 to 12.50]

4. Primary Outcome: Change in Brown Spots at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of spots
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of spots
  Front | -0.50 [-12.00 to 9.00]
  Left Oblique | -4.00 [-9.50 to 6.50]
  Nose | -0.50 [-3.50 to 1.50]
  Right Oblique | 8.50 [-14.00 to 22.50]

5. Primary Outcome: Change in Pores at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall pore count using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement.
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of pores
Groups:
- Single Treatment Arm: Quantitively assessment of pore count using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of pores
  Front | -5.00 [-11.00 to 10.00]
  Left Oblique | -5.00 [-13.00 to 17.00]
  Nose | -11.00 [-21.00 to 3.00]
  Right Oblique | -3.00 [-7.00 to 10.00]

6. Primary Outcome: Change in Pores at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 5
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of pores
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of pores
  Front | 1.00 [-34.00 to 14.00]
  Left Oblique | -1.00 [-6.00 to 17.00]
  Nose | 1.00 [-15.00 to 5.00]
  Right Oblique | -7.00 [-21.00 to 3.00]

7. Primary Outcome: Change in Pores at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 5
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of pores
Groups:
- Double Treatment Arm: Quantitively assessment of pore count using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of pores
  Front | 2.50 [-41.00 to 23.50]
  Left Oblique | -27.50 [-72.00 to 10.00]
  Nose | -10.00 [-28.00 to -5.50]
  Right Oblique | -17.00 [-60.00 to 34.00]

8. Primary Outcome: Change in Pores at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 5
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of pores
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of pores
  Front | -0.00 [-0.00 to -0.00]
  Left Oblique | -0.00 [-0.00 to 0.00]
  Nose | -0.00 [-0.01 to 0.00]
  Right Oblique | -0.00 [-0.00 to 0.00]

9. Primary Outcome: Change in Porphyrins at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall porphyrins count using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement.
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of porphyrins
Groups:
- Single Treatment Arm: Quantitively assessment of porphyrins count using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of porphyrins
  Front | 17.00 [-292.00 to 217.00]
  Left Oblique | 51.00 [-381.00 to 331.00]
  Nose | 15.00 [-49.00 to 66.00]
  Right Oblique | 4.00 [-290.00 to 351.00]

10. Primary Outcome: Change in Porphyrins at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 9
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of porphyrins
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of porphyrins
  Front | -123.00 [-365.00 to 272.00]
  Left Oblique | -192.00 [-446.00 to 99.00]
  Nose | 32.00 [-19.00 to 88.00]
  Right Oblique | -114.00 [-420.00 to 136.00]

11. Primary Outcome: Change in Porphyrins at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 9
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of porphyrins
Groups:
- Double Treatment Arm: Quantitively assessment of porphyrins count using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of porphyrins
  Front | 1.00 [-312.00 to 395.50]
  Left Oblique | 164.50 [-56.50 to 730.00]
  Nose | 45.50 [-25.00 to 94.50]
  Right Oblique | 214.50 [-39.50 to 789.50]

12. Primary Outcome: Change in Porphyrins at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 9
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of porphyrins
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of porphyrins
  Front | -160.50 [-266.00 to -1.00]
  Left Oblique | -145.50 [-263.00 to 158.50]
  Nose | 3.00 [-66.00 to 60.00]
  Right Oblique | 13.00 [-278.50 to 135.50]

13. Primary Outcome: Change in Red Features at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall red features using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement
Time Frame: Baseline, 1 Month
Population: Analysis was focused on testing whether the effect of the treatment on each parameter differed Frontal- 2 subjects data was incomplete. Left- 1 subject data was incomplete
  The per-protocol (PP) population will be the primary population for all statistical analyses. The PP population will include all subjects who received treatment and completed the study in general accordance with the protocol. Only the data of completing subjects will be analyzed.
Measure: Median (Inter-Quartile Range); unit: count of red features
Groups:
- Single Treatment Arm: Quantitively assessment of intensity in overall red areas using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of red features
  Front: number analyzed (Participants) | 5
  Front | 1.00 [-1.00 to 5.00]
  Left Oblique: number analyzed (Participants) | 6
  Left Oblique | -7.00 [-10.00 to 2.00]
  Nose | -1.00 [-3.00 to 10.00]
  Right Oblique | -2.00 [-7.00 to 12.00]

14. Primary Outcome: Change in Red Features at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 13
Time Frame: Baseline, 3 Months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: count of red features
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of red features
  Front: number analyzed (Participants) | 5
  Front | 2.00 [-6.00 to 5.00]
  Left Oblique: number analyzed (Participants) | 6
  Left Oblique | -7.00 [-12.00 to 7.00]
  Nose | 0.00 [-4.00 to 3.00]
  Right Oblique | 0.00 [-17.00 to 9.00]

15. Primary Outcome: Change in Red Features at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 13
Time Frame: Baseline, 1 Month
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: count of red features
Groups:
- Double Treatment Arm: Quantitively assessment of intensity in overall red areas using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of red features
  Front: number analyzed (Participants) | 6
  Front | 4.00 [1.50 to 9.00]
  Left Oblique: number analyzed (Participants) | 7
  Left Oblique | 7.50 [-1.50 to 11.00]
  Nose | 0.00 [-2.50 to 2.50]
  Right Oblique | 3.50 [-14.00 to 8.50]

16. Primary Outcome: Change in Red Features at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 13
Time Frame: Baseline, 3 Months
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: count of red features
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of red features
  Front: number analyzed (Participants) | 6
  Front | 2.00 [-0.50 to 9.50]
  Left Oblique: number analyzed (Participants) | 7
  Left Oblique | 5.50 [1.00 to 15.00]
  Nose | 1.00 [-2.00 to 3.00]
  Right Oblique | 2.50 [-10.50 to 5.00]

17. Primary Outcome: Change in Texture at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall texture using measurements provided VISIA 3D analysis on different sides of the face for all subjects. Skin analysis is performed by the system to generate a numerical roughness count by providing a tally of the feature.
  A lower value signifies improvement. Minimum and Maximum value does not exist.
  The value is an Absolute Score derived from the integration of multiple topographical variables; because it measures the intensity of texture rather than a specific length or depth, it has no standard metric unit
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: unitless
Groups:
- Single Treatment Arm: Quantitively assessment of intensity in overall texture using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
unitless
  Front | -14.00 [-125.00 to 521.00]
  Left Oblique | -3.00 [-336.00 to 354]
  Nose | -1.00 [-42.00 to 14.00]
  Right Oblique | 68.00 [-99.00 to 453.00]

18. Primary Outcome: Change in Texture at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 17
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: unitless
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
unitless
  Front | 64.00 [-210.00 to 147.00]
  Left Oblique | 188.00 [45.00 to 302.00]
  Nose | 30.00 [-30.00 to 302.00]
  Right Oblique | 161.00 [19.00 to 396.00]

19. Primary Outcome: Change in Texture at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 17
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: unitless
Groups:
- Double Treatment Arm: Quantitively assessment of intensity in overall texture using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
unitless
  Front | 20.50 [-216.00 to 413.00]
  Left Oblique | -198.00 [-569.00 to 155.00]
  Nose | 4.00 [-19.00 to 41.50]
  Right Oblique | -225.50 [-506.00 to -25.00]

20. Primary Outcome: Change in Texture at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 17
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: unitless
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
unitless
  Front | -25.00 [-146.50 to 212.50]
  Left Oblique | 82.00 [-141.00 to 236.00]
  Nose | 16.50 [-2.50 to 43.00]
  Right Oblique | -72.00 [-246.00 to 171.00]

21. Primary Outcome: Change in UV Spots at 1 Month From Baseline (Single Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of UV spots
Groups:
- Single Treatment Arm: Quantitively assessment of intensity in overall uv spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of UV spots
  Front | -4.00 [-8.00 to -1.00]
  Left Oblique | -4.00 [-11.00 to 3.00]
  Nose | 0.00 [-6.00 to 2.00]
  Right Oblique | 0.00 [-1.00 to 11.00]

22. Primary Outcome: Change in UV Spots at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of UV spots
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of UV spots
  Front | -3.00 [-15.00 to 6.00]
  Left Oblique | -4.00 [-12.00 to 11.00]
  Nose | -2.00 [-3.00 to 1.00]
  Right Oblique | 1.00 [-4.00 to 3.00]

23. Primary Outcome: Change in UV Spots at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of UV spots
Groups:
- Double Treatment Group: Quantitively assessment of intensity in overall uv spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Group
Number analyzed (Participants) | 8
count of UV spots
  Front | -1.50 [-11.50 to 7.50]
  Left Oblique | 5.00 [-19.50 to 11.50]
  Nose | -2.50 [-5.50 to 1.00]
  Right Oblique | -1.00 [-25.00 to 6.00]

24. Primary Outcome: Change in UV Spots at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 1
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of UV spots
Groups:
- Double Treatment Arm: Quantitively assessment of intensity in overall uv spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of UV spots
  Front | -1.00 [-15.00 to 4.50]
  Left Oblique | -7.50 [-15.50 to 13.50]
  Nose | -2.50 [-4.00 to 1.00]
  Right Oblique | 4.50 [-7.50 to 10.50]

25. Primary Outcome: Change in Visible Spots at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall visible spots using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of visible spots
Groups:
- Single Treatment Arm: Subjects received a single treatment of BBL, HALO and MOXI.
  Quantitively assessment of intensity in overall visible spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of visible spots
  Frontal | 2.00 [0.00 to 12.00]
  Left Oblique | -3.00 [-6.00 to 4.00]
  Nose | -1.00 [-1.00 to 0.00]
  Right Oblique | 3.00 [1.00 to 5.00]

26. Primary Outcome: Change in Visible Spots at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 25
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of visible spots
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
count of visible spots
  Frontal | 6.00 [3.00 to 9.00]
  Left Oblique | 1.00 [-3.00 to 4.00]
  Nose | 0.00 [-1.00 to 5.00]
  Right Oblique | 3.00 [-4.00 to 3.00]

27. Primary Outcome: Change in Visible Spots at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 25
Time Frame: Baseline, 1 Month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of visible spots
Groups:
- Double Treatment Arm: Subjects received a single treatment of BBL, HALO and MOXI.
  Quantitively assessment of intensity in overall visible spots using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of visible spots
  Frontal | 6.00 [-12.50 to 20.50]
  Left Oblique | -6.50 [-11.50 to 6.50]
  Nose | -0.50 [-2.50 to 0.50]
  Right Oblique | -11.00 [-14.00 to 6.00]

28. Primary Outcome: Change in Visible Spots at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 25
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: count of visible spots
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
count of visible spots
  Frontal | -2.00 [-5.00 to 4.00]
  Left Oblique | 0.00 [-7.50 to 8.50]
  Nose | -0.50 [-1.00 to 1.50]
  Right Oblique | -0.50 [-5.50 to 11.00]

29. Primary Outcome: Change in Total Wrinkle Area at 1 Month From Baseline (Single Treatment Group)
Description: Quantitively assessment of change in overall wrinkle are using measurements provided VISIA 3D analysis on different sides of the face for all subjects
  A lower value signifies improvement.
Time Frame: Baseline, 1 Month
Population: Analysis was focused on testing whether the effect of the treatment on each parameter differed Nose- 1 subject didn't have complete data thus it was not included in analysis
  The per-protocol (PP) population will be the primary population for all statistical analyses. The PP population will include all subjects who received treatment and completed the study in general accordance with the protocol. Only the data of completing subjects will be analyzed.
Measure: Median (Inter-Quartile Range); unit: mm^2
Groups:
- Single Treatment Arm: Quantitively assessment of wrinkle area using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
mm^2
  Front | -1.00 [-3.00 to 0.00]
  Left Oblique | -13.00 [-17.00 to -3.00]
  Nose: number analyzed (Participants) | 6
  Nose | -3.00 [-3.00 to 0.00]
  Right Oblique | 5.00 [-63.00 to 12.00]

30. Primary Outcome: Change in Total Wrinkle Area at 3 Months From Baseline (Single Treatment Group)
Description: as for outcome 29
Time Frame: Baseline, 3 Months
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 7
mm^2
  Front | -1.00 [-2.00 to 3.00]
  Left Oblique | -1.00 [-12.00 to 18.00]
  Nose: number analyzed (Participants) | 6
  Nose | 1.00 [-5.00 to 1.00]
  Right Oblique | 5.00 [-24.00 to 24.00]

31. Primary Outcome: Change in Total Wrinkle Area at 1 Month From Baseline (Double Treatment Group)
Description: as for outcome 29
Time Frame: Baseline, 1 Month
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: mm^2
Groups:
- Double Treatment Arm: Quantitively assessment of wrinkle area using measurements provided from VISIA 3D analysis
  A lower value signifies improvement
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
mm^2
  Front | 0.50 [-3.00 to 1.00]
  Left Oblique | -14.50 [-42.00 to 0.50]
  Nose: number analyzed (Participants) | 7
  Nose | -2.50 [-5.50 to -0.50]
  Right Oblique | -14.50 [-39.50 to -2.00]

32. Primary Outcome: Change in Total Wrinkle Area at 3 Months From Baseline (Double Treatment Group)
Description: as for outcome 29
Time Frame: Baseline, 3 Months
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: mm^2
Arm/Group | Double Treatment Arm
Number analyzed (Participants) | 8
mm^2
  Front | 0.00 [-2.00 to 0.00]
  Left Oblique | 12.00 [-16.00 to 21.50]
  Nose: number analyzed (Participants) | 7
  Nose | -1.00 [-4.50 to 2.50]
  Right Oblique | -13.50 [-31.50 to 6.00]

ADVERSE EVENTS:
Time Frame: 4 months
Description: similar treatment parameters allowed for overall assessment
Groups:
- Single Treatment Group Participants: all reportable events for all patients who underwent single treatment (1 BBL/MOXI/HALO treatments)
- Double Treatment Group Participants: all reportable events for all patients who underwent double treatment (2 BBL/MOXI/HALO treatments)
Arm/Group | Single Treatment Group Participants | Double Treatment Group Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT06091215/Prot_SAP_000.pdf